CLINICAL TRIAL: NCT00015457
Title: Trial of Amlodipine Combined With Botulinum Toxin Injections for Focal Dystonia
Brief Title: Amlodipine Plus Botulinum Toxin for Focal Dystonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Barbara Karp, M.D., MD, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 010147; 01-N-0147 (Other: NIH)
Record Dates: First submitted 2001-04-18; First posted 2001-04-19 (Estimated); Results first posted 2013-04-01 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2013-03

CONDITIONS: Focal Dystonia
Keywords: Writer's Cramp; Calcium Channel Antagonists; Torticollis; Chemodenervation
MeSH Terms: conditions — Dystonic Disorders; Torticollis | interventions — Amlodipine; Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (1):
- cervical dystonia (Experimental): cervical dsytonia patinets
  Interventions: Drug: Amlodipine plus Botulinum toxin

INTERVENTIONS:
Drug: Amlodipine plus Botulinum toxin

SUMMARY:
Objective: To determine if the calcium channel blockers, amlodipine can augment the effect of botulinum toxin injections in the treatment of focal dystonia.

Study Population: 20 patients with cervical dystonia

Design: Double-bind, placebo-controlled clinical trail.

Outcome measures: For patients: dystonia rating scales (Twistrs, Fahn-Marsden dystonia scale, NINDS subjective patient rating scale), and hand grip strength. For healthy volunteers: Amplitude of EDB MEP.

DETAILED DESCRIPTION:
Objective: To determine if the calcium channel blocker, amlodipine can augment the effect of botulinum toxin injections in the treatment of focal dystonia.

Study Population: 20 patients with cervical dystonia

Design: Double-bind, placebo-controlled clinical trail.

Outcome measures: dystonia rating scales (TWISTRS)

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients enrolled in Protocol 85-N-0195, Efficacy and Pathophysiology of Botulinum Toxin for Treatment of Involuntary Movement Disorders are eligible for enrollment if they meet the following inclusion and exclusion criteria.

Good general health

Focal hand dystonia or cervical dystonia

Stable response to botulinum toxin demonstrated through a series of at least 3 injections over a period of at least a year

Benefit from the 3 immediately prior btx injections rated as 75% or less or a duration of benefit lasting less than or equal to 2 months

No other medications for dystonia

EXCLUSION CRITERIA:

Cervical dystonia accompanied by dysphagia or dyspnea, either before or with botulinum toxin injection

Present or past cardiac disease, hypertension, arrhythmia or congestive heart failure

Anterocollis or other neck dystonia requiring bilateral anterior neck muscle injections

Use of concomitant medications affecting calcium channels or those metabolized by the cytochrome p450 3A4 system including grapefruit juice, St. John's wort, HIV protease inhibitors, cimetidine, antibiotics (macrolides, fluoroquinones, antifungal, rifampin), antidepressants (fluvoxamine, norfluoxetine), barbiturates, anticonvulsants (carbamazepine, phenytoin), oral diabetes agents (pioglitazone, troglitazone), and glucocorticoids

Allergy to amlodipine or related compounds

Pregnany/ nursing

Age less than 18 years of age

Abnormal EKG

Abnormal coagulation profile or liver function tests

Use of anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2001-04; Primary Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anderson RL, Patel BC, Holds JB, Jordan DR. Blepharospasm: past, present, and future. Ophthalmic Plast Reconstr Surg. 1998 Sep;14(5):305-17. PMID 9783280
- [Background] Jankovic J, Schwartz K. Botulinum toxin injections for cervical dystonia. Neurology. 1990 Feb;40(2):277-80. doi: 10.1212/wnl.40.2.277. PMID 2300249
- [Background] Jankovic J, Schwartz K, Donovan DT. Botulinum toxin treatment of cranial-cervical dystonia, spasmodic dysphonia, other focal dystonias and hemifacial spasm. J Neurol Neurosurg Psychiatry. 1990 Aug;53(8):633-9. doi: 10.1136/jnnp.53.8.633. PMID 2213039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from a medical clinic providing botulinum toxin treatment for cervical dystonia. Patients recruited between 6/21/01 and 10/19/06
Pre-assignment Details: Patients were excluded if response to previous btx injections were not stable, serious medical conditions, pregnancy, abnormal medical screening
Groups:
- Amlodipine Then Placebo: Patients with cervical dystonia receiving botulinum toxin injections plus Amlodipine during the first period and botulinum toxin injections plus Placebo during the second period.
- Placebo Then Amlodipine: Patients with cervical dystonia receiving botulinum toxin injections plus Placebo during the first period and botulinum toxin injections plus Amlodipine during the second period.
Period: First Intervention
Arm/Group | Amlodipine Then Placebo | Placebo Then Amlodipine
Started | 8 | 8
Completed | 8 | 5
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 0 | 1
Period: Second Intervention
Arm/Group | Amlodipine Then Placebo | Placebo Then Amlodipine
Started | 8 | 5
Completed | 7 | 5
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cervical Dystonia: All participants enrolled in study
Arm/Group | Cervical Dystonia
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants] — age >18
  Participants
    <=18 years | 0
    Between 18 and 65 years | 15
    >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Toronto Western Spasmodic Torticollis Rating Scale (TWSTR) Sum Score
Description: Rating scale assessing sum of severity of dystonia, disability score and pain scale. Ordinal scale ranging from 0 (least severe) to 30 (maximally severe). Score is maximal response TWSTR rating minus baseline rating.
Time Frame: 1-2 month maximal rating
Population: Total enrolled less withdrawals from study. One participant completed the study but did not yield analyzeable data
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Amlodipine: Patients receiving Amlodipine plus botulinum toxin injections during either period.
- Placebo: Patients receiving Placebo plus botulinum toxin injections during either period.
Arm/Group | Amlodipine | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale | -6.00 (10.23) | -3.23 (6.06)

2. Secondary Outcome: Duration of Response to Botulinum Toxin Injection With Amlodipine and With Placebo
Description: Self reported duration of effect in weeks.
Time Frame: 3 months
Population: Total enrolled less withdrawals. Less one participant who completed the study but who did not yield analyzeable data.
Measure: Median (Full Range); unit: weeks
Arm/Group | Amlodipine | Placebo
Number analyzed (Participants) | 11 | 11
weeks | 6 [1 to 12] | 5.5 [2 to 12]

ADVERSE EVENTS:
Arm/Group | Amlodipine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amlodipine (N=16) | Placebo (N=16)
hypereosinophila (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
dysphagia (General disorders) | 0 (0) | 1 (1)
swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — ankle edema

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes